CLINICAL TRIAL: NCT05663242
Title: To Compare the Effects of Intraoperative Use of Intravenous Anesthetics Propofol and Inhaled Anesthetics Sevoflurane on the Prognosis of Patients Undergoing Surgery for Primary Lung Tumors and the Investigation of Its Mechanism of Action.
Brief Title: The Effects of Using Different Anesthetics on the Prognosis of Primary Lung Tumors and Its Mechanism of Action
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210218.
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer; Progression, Disease; Anesthesia
Keywords: Propofol; Sevoflurane; Lung Cancer; VATS
MeSH Terms: conditions — Lung Neoplasms; Disease Progression | interventions — Propofol; Sevoflurane; Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Experimental): The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3).
  Interventions: Drug: Sevoflurane
- Propofol (Experimental): The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Other Names: total intravenous anesthesia
  Arms: Propofol
Drug: Sevoflurane — The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3 MAC)
  Other Names: inhalation anesthesia
  Arms: Sevoflurane

SUMMARY:
This is a two-arm, parallel-group randomized clinical trial. Routine perioperative care would be performed in volunteers with primary early lung cancer. The study will enroll approximately 300 volunteers to compare the progression-free or overall survival in patients undergoing video-assisted thoracoscopic surgery (VATS) for primary lung tumors between propofol and sevoflurane for the maintenance of anesthesia.

DETAILED DESCRIPTION:
Before the scheduled procedure, the patients are randomly assigned into peopofol group or groups (1:1) according to the randomization generated by the computer. Both groups were induced with propofol 1~2.5 mg/kg propofol. The propofol group was maintained at an effect-site concentration of 2.0-4.0 mcg/mL by a target-controlled infusion system. The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3 MAC). During the operation, the dose of anesthetic drugs (propofol/fentanyl /remifentanil and sevoflurane/cisatracurium/rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value and Entropy (or BIS) value at 40-60in both groups. The following patient data were recorded, the type of anesthesia, sex, age at the time of surgery, preoperative Karnofsky performance status score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), American Society of Anesthesiologists physical status scores, tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/fentanyl/ propofol) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, and 3-year overall survival and Karnofsky performance status score were recorded.

ELIGIBILITY:
Inclusion Criteria:

* eighteen to eighty-year-old
* ASA class I-III patients
* Received elective thoracic surgery for primary lung tumors under general anesthesia

Exclusion Criteria:

* mental disorder
* poor liver function
* pregnant or lactating women
* morbidly obese
* allergy to any of the drugs used in this study
* recurrent tumor or repeat surgery
* biopsy cases
* incomplete outcome-data
* palliative treatment after surgery
* simultaneous treatment of other malignancies
* emergency surgery
* presence of other malignant tumors
* combined propofol and inhalation anesthesia or other anesthetics, such as ketamine or dexmedetomidine
* diagnosed as benign lung tumor, or other metastatic lung tumor

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  6-month overall survival, 1-year overall survival, and 3-year overall survival
The presence of disease progression | From the date of surgery until the date of first documented progression (recurrence or metastasis),assessed up to 36 months
  From the date of surgery until the date of first documented progression (recurrence or metastasis) or date of death from any cause, assessed up to 36 months

SECONDARY OUTCOMES:
Postoperative complications | The period from the day of surgery to postoperative 30 days
  Clavien-Dindo classification, and other postoperative complications
Karnofsky performance status score | Karnofsky performance score(from 0 (dead) to 100(normal no complication)) before surgery (baseline data) , postoperation 7 days, postoperation 3 months, postoperation 6 months, postoperation 12 months
  to access patients' functional impairment
Length of hospital stays | from the day of surgery to dischage, assessed up to 30 days
  the length of stays in general ward and ICU

OTHER OUTCOMES:
time of operation and anesthesia | time of the total procedure
  record the time the opeartion and anesthesia
blood loss | during the operation of VATS
  record the blood loss (ml)
volume of blood transfusion | during the operation of VATS
  volume of blood transfusion (ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan